CLINICAL TRIAL: NCT06628492
Title: Comparative Assessment for the Positional Accuracy of Dental Implants Inserted by Computerized Surgical Guides Fabricated From Different Printing Materials
Brief Title: Surgical Guided Fabricated From Two Different Printing Materials
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 802/2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A implant inserted by stainless steel surgical guide (Experimental)
  Interventions: Device: stainless steel printed surgical guide
- group B implant inserted by resin surgical guide (Active Comparator)
  Interventions: Device: resin printed surgical guide

INTERVENTIONS:
Device: stainless steel printed surgical guide — the patient will wear the stainless steel surgical guide for the insertion of one implant
  Arms: group A implant inserted by stainless steel surgical guide
Device: resin printed surgical guide — the patient will wear the resin surgical guide for insertion of adjacent another implant implant
  Arms: group B implant inserted by resin surgical guide

SUMMARY:
implant will be inserted in patients with kennedy class 3 or 4 partially edentulous mandible .the implants will be inserted using teeth supported surgical guide fabricated from two different materials

ELIGIBILITY:
Inclusion Criteria:

1. Patients with skeletal Angle´s class I maxilla-mandibular relationship,
2. adequate inter-arch distance, have Kennedy class 3 or 4 partially edentulous mandible of more than 2 teeth missed and will be applied for the treatment of tooth loss and requiring fixed prosthodontic rehabilitation
3. normal Physical and psychological status to tolerate conventional implant procedures,
4. Their residual ridge had sufficient bone volume for implant installation and was covered by firm mucoperiosteum.

Exclusion Criteria:

1. Smokers.
2. Patients undergoing chemotherapy or radiotherapy and immunocompromised patients.
3. Patients with, systemic disease that might complicate post-operative healing or contribute to bone resorption, e.g uncontrolled diabetes, psychological disorders, or alcohol, tobacco, or drug abuse
4. parafunctional habits, poor oral hygiene, limited mouth opening, severe alveolar bone deficiencies,

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
linear deviation of inserted implant | 1 month
  coronal and apical deviation of inserted implant from virtually planned one in millimeter.
angular deviation of inserted implant | 1 month
  angular deviation of inserted implant from virtually planned one in angles.